CLINICAL TRIAL: NCT00006482
Title: A Phase II Evaluation Of Gemcitabine And Cisplatin In Persistent Or Recurrent Squamous Cell Carcinoma Of The Cervix
Brief Title: Gemcitabine and Cisplatin in Treating Patients With Refractory or Recurrent Cancer of the Cervix
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000068313; GOG-0127Q
Record Dates: First submitted 2000-11-06; First posted 2003-10-08 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2004-05

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; stage IVB cervical cancer; stage IVA cervical cancer; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Gemcitabine

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine and cisplatin in treating patients who have refractory or recurrent cancer of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of gemcitabine and cisplatin in patients with refractory or recurrent squamous cell carcinoma of the cervix.
* Determine the nature and degree of toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive cisplatin IV and gemcitabine IV over 1 hour on days 1 and 8. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 28-69 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed refractory or recurrent squamous cell carcinoma of the cervix that has failed local therapy and is considered incurable
* Must have had 1 prior chemotherapy regimen for cervical cancer

  * No more than 1 prior chemotherapy regimen (single or combination drug therapy), unless used as a radiosensitizer
  * No prior chemotherapy for recurrent or persistent disease including retreatment with initial chemotherapy
* Bidimensionally measurable disease
* Ineligible for higher priority GOG protocol

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least lower limit of normal
* Absolute neutrophil count at least 1,500/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT and alkaline phosphatase no greater than 3 times normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* Not pregnant
* Fertile patients must use effective contraception
* No significant infection
* No other malignancies within past 5 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 3 weeks since prior biologic therapy for cervical cancer

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy for cervical cancer and recovered
* No prior gemcitabine

Endocrine therapy:

* At least 3 weeks since prior endocrine therapy for cervical cancer

Radiotherapy:

* At least 3 weeks since prior radiotherapy for cervical cancer and recovered
* No prior radiotherapy to more than 25% of marrow-bearing areas

Surgery:

* At least 3 weeks since prior surgery for cervical cancer and recovered

Other:

* No concurrent amifostine or other protective reagents
* No prior anticancer therapy that contraindicates study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-10; Primary Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A. Brewer, MD, Study Chair — University of Illinois College of Medicine at Peoria
Locations (34):
- United States (33):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Rational Therapeutics Inc., Long Beach, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Illinois College of Medicine at Peoria, Peoria, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Tufts University School of Medicine, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital at North Shore, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - Tacoma General Hospital, Tacoma, Washington
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Brewer CA, Blessing JA, Nagourney RA, McMeekin DS, Lele S, Zweizig SL. Cisplatin plus gemcitabine in previously treated squamous cell carcinoma of the cervix: a phase II study of the Gynecologic Oncology Group. Gynecol Oncol. 2006 Feb;100(2):385-8. doi: 10.1016/j.ygyno.2005.09.009. Epub 2005 Nov 4. PMID 16271750